CLINICAL TRIAL: NCT04674644
Title: Suleyman Demirel University Faculty of Dentistry Pediatric Dentistry Department
Brief Title: Analysing the Psychosocial Effects of COVID-19 Pandemic on Dental Professionals Using the Turkish Version of the Fear of COVID-19 and Coronavirus Anxiety Scales
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Esra Oz, Assistant Professor, Suleyman Demirel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 355
Record Dates: First submitted 2020-12-16; First posted 2020-12-19 (Actual); Results first posted 2021-01-29 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: COVID-19 Pandemic
Keywords: Fear of COVID-19; Coronavirus anxiety scale; COVID-19; dental professionals; psychosocial effects
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Dental professionals
Masking Description: Dental professionals working in public and university hospitals
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Analysing the psychosocial effects of COVID-19 pandemic on dental professionals (Other): Dental professionals
  Interventions: Behavioral: The psychosocial effects of COVID-19 pandemic on dental professionals

INTERVENTIONS:
Behavioral: The psychosocial effects of COVID-19 pandemic on dental professionals — Analysing the psychosocial effects of COVID-19 pandemic on dental professionals using the Turkish version of the Fear of COVID-19 and Coronavirus Anxiety Scales

SUMMARY:
The aims of this study were to (i) assess fear and anxiety of COVID-19 in a Turkish sample dental professionals using the Turkish FCV-19S and CAS; (ii) explore factors associated with FCV-19S and CAS; and (iii) examine the psychometric properties of the Turkish FCV-19S and CAS.

DETAILED DESCRIPTION:
This cross-sectional study was conducted between October, 16 to 23, 2020 by sending an online survey questionnaire working in public and university hospitals, including general dentists or specialists. The tool utilized for data collection was a designed online Google Forms questionnaire.

This survey was implemented by using a questionnaire that included socio-demographic data (age range, gender, marital status, systemic disease, professional area, years of clinical experience, number of patients treated daily, smoking status, alcohol consumption, vs), epidemic-related questions and scales measuring the fear and anxiety levels of the participants.

Fear of COVID-19 Scale is an unidimensional scale seven-item scale assessing anxiety regarding COVID-19 developed by Ahorsu et al. Items are rated on a 5-item Likert scale from 1 (Strongly disagree) to 5 (Strongly agree) with scores ranging from 7 to 35. A higher score of the FCV-19S represents a greater level of fear. In the study, the bi-factor model and two-factor model consisting of the "emotional response" factor (items 1, 2, 4, and 5) and "physiological response" factor (items 3, 6, and 7) were used.

Coronavirus Anxiety Scale is an unidimensional tool that assesses the physiological reactions anxiety related to the COVID-19 pandemic. Participants were asked to rate 5 items on a 5-point Likert-type scale, from 0 (not at all) to 4 (nearly every day over the last 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Dental professionals working in public hospitals
* Dental professionals working in university hospitals

Exclusion Criteria:

* Dental professionals working in private clinics

Min Age: 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: esra Oz, Assist Prof, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University Faculty of Dentistry Pediatric Dentistry Department, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahmood QK, Jafree SR, Qureshi WA. The Psychometric Validation of FCV19S in Urdu and Socio-Demographic Association with Fear in the People of the Khyber Pakhtunkhwa (KPK) Province in Pakistan. Int J Ment Health Addict. 2022;20(1):426-436. doi: 10.1007/s11469-020-00371-4. Epub 2020 Jul 12. PMID 32837443
- [Background] Ahmed O, Faisal RA, Sharker T, Lee SA, Jobe MC. Adaptation of the Bangla Version of the COVID-19 Anxiety Scale. Int J Ment Health Addict. 2022;20(1):284-295. doi: 10.1007/s11469-020-00357-2. Epub 2020 Jun 27. PMID 32837436
- [Background] Alyami M, Henning M, Krageloh CU, Alyami H. Psychometric Evaluation of the Arabic Version of the Fear of COVID-19 Scale. Int J Ment Health Addict. 2021;19(6):2219-2232. doi: 10.1007/s11469-020-00316-x. Epub 2020 May 16. PMID 32427217
- [Background] Andrade EF, Pereira LJ, Oliveira APL, Orlando DR, Alves DAG, Guilarducci JS, Castelo PM. Perceived fear of COVID-19 infection according to sex, age and occupational risk using the Brazilian version of the Fear of COVID-19 Scale. Death Stud. 2022;46(3):533-542. doi: 10.1080/07481187.2020.1809786. Epub 2020 Aug 26. PMID 32845795

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with missing data were excluded from the study
Groups:
- Analysing the Psychosocial Effects of COVID-19 Pandemic: General dentists and specialists analyzed during COVID-19 pandemic
Period: Overall Study
Arm/Group | Analysing the Psychosocial Effects of COVID-19 Pandemic
Started (number of participants) | 850
Completed (number of participants) | 813
Not Completed | 37
Not completed — with missing data | 37

BASELINE CHARACTERISTICS:
Groups:
- Analysing the Psychosocial Effects of COVID-19 Pandemic on Dental Professionals: Data were collected by sending an online survey questionnaire to dentists working in public and university hospitals, including both general dentists and specialists.
  The survey consisted of a questionnaire that included sociodemographic data (age range, gender, marital status, composition of household, systemic disease, professional area, years of clinical experience, number of patients treated daily, smoking status, alcohol consumption), epidemic-related questions, and scales measuring the fear and anxiety levels of the participants. In the last part of the survey, the levels of fear and anxiety were assessed by the FCV-19S and CAS.
Arm/Group | Analysing the Psychosocial Effects of COVID-19 Pandemic on Dental Professionals
Number analyzed (Participants) | 813
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 813
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 30 [23 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 553
  Male | 260
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 813
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 813

OUTCOME MEASURES:

1. Primary Outcome: The Psychosocial Effects of COVID-19 Pandemic on Dental Professionals Using the Turkish Version of the Fear of COVID-19 Scale
Description: Fear of COVID-19 Scale is an unidimensional scale seven-item scale assessing anxiety regarding COVID-19 . Items are rated on a 5-item Likert scale from 1 (Strongly disagree) to 5 (Strongly agree) with scores ranging from 7 to 35. Scores are added up. A higher score of the FCV-19S represents a greater level of fear and a worse outcome.
Time Frame: during the survey administration
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Analysing the Psychosocial Effects of COVID-19 Pandemic on Dental Professionals: General dentists and specialists
Arm/Group | Analysing the Psychosocial Effects of COVID-19 Pandemic on Dental Professionals
Number analyzed (Participants) | 813
scores on a scale | 18.48 (5.47)

2. Secondary Outcome: The Psychosocial Effects of COVID-19 Pandemic Using the Turkish Version of the Coronavirus Anxiety Scale
Description: Coronavirus Anxiety Scale is an unidimensional tool that assesses the physiological anxiety related to the COVID-19. Participants rated 5 items on a 5-point Likert-type scale, from 0 (not at all) to 4 (nearly every day over the last 2 weeks). Scores are added up for a total score of 0 - 20, with higher scores indicating worse outcomes.
Time Frame: during the survey administration
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- The Psychosocial Effects of COVID-19 Using the Turkish Version of the Coronavirus Anxiety Scale: General dentists and specialists
Arm/Group | The Psychosocial Effects of COVID-19 Using the Turkish Version of the Coronavirus Anxiety Scale
Number analyzed (Participants) | 813
scores on a scale | 2.17 (3.08)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Groups:
- Analysing the Psychosocial Effects of COVID-19 Pandemic on Dental Professionals: The psychosocial effects of COVID-19 pandemic on general dentists and specialists
Arm/Group | Analysing the Psychosocial Effects of COVID-19 Pandemic on Dental Professionals
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The present study has some limitations. Since the stress and anxiety levels of the dentists participating in the study prior to the pandemic are not known, the extent of the increase in these levels is unknown. In addition, because this is a cross-sectional study, the findings reflect only a certain period of the pandemic. Only scales related to COVID-19 were included, as it was thought that participants might be reluctant to participate in a longer survey.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT04674644/Prot_SAP_000.pdf